CLINICAL TRIAL: NCT04370015
Title: Efficacy and Safety of Hydroxychloroquine in Primary Prophylaxis of SARS-CoV-2 Infection in Healthcare Workers at Risk of Exposure: Randomised Control Trial
Brief Title: Hydroxychloroquine Chemoprophylaxis for COVID-19 Infection in High-risk Healthcare Workers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr. Saira Burney, Doctor, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16082019
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2; Healthcare Workers
Keywords: SARS-CoV-2; HCQ; prophylaxis; healthcare workers
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Health care workers at high risk of contracting SARS-CoV-2 randomized to this arm will be treated with oral hydroxychloroquine 400 mg twice a day (four 200 mg tablets) on day 1 followed by 400mg (two 200 mg tablets) once a week for 11 weeks.
  Interventions: Drug: Hydroxychloroquine
- Control group (Placebo Comparator): Health care workers at high risk of contracting SARS-CoV-2 randomized to this arm will be treated with placebo twice a day (four tablets) on day 1 followed by 2 tablets once a week for 11weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — Health care workers at high risk of contracting SARS-CoV-2 randomized to this arm will be treated with oral hydroxychloroquine 400 mg twice a day (four 200 mg tablets) on day 1 followed by 400mg (two 200 mg tablets) once a week for 11 weeks.
  Other Names: HCQ
  Arms: Treatment group
Drug: Placebo oral tablet — • Health care workers at high risk of contracting SARS-CoV-2 randomized to this arm will be treated with placebo twice a day (four tablets) on day 1 followed by 2 tablets once a week for 11weeks.
  Arms: Control group

SUMMARY:
Healthcare personnel are at an increased risk of exposure to SARS-CoV-2 infection while handling such patients. Currently, there is no treatment available for SARS-CoV-2 and stringent preventive measures are advised to avoid or minimize risk of exposure to healthcare workers. There are in vitro studies available which show inhibition of corona virus by hydroxychloroquine, a widely-used agent against malaria and certain autoimmune conditions and of low-cost and limited toxicity. However, evidence regarding its effects in patients is limited. We plan to conduct a randomized controlled trial to evaluate the safety and potential prophylactic efficacy of hydroxychloroquine in preventing secondary SARS-CoV-2 infection among healthcare workers at high-risk of exposure while managing such patients.

DETAILED DESCRIPTION:
An interventional randomised control trial that will include 374 participants who will be healthcare workers at variable risks of exposure to SARS-CoV-2 while managing patients both suspected and confirmed with COVID-19 infection.Each participant will undergo detailed clinical evaluation to confirm eligibility, complete blood count, retinal imaging and ECG rhythm lead at baseline. A nasopharyngeal swab for reverse-transcriptase-polymerase chain reaction (RT-PCR) will also be taken. The enrolled participants will be randomised to two treatment arms with the experimental arm receiving Tab.Hydroxychloroquine (HCQ) 400mg twice a day on day 1 followed by 400mg weekly for 11 weeks. The placebo comparator arm will receive 2 tablets twice daily on day 1 followed by 2 tablets weekly for 11 weeks. The participants will be followed up via phone call weekly to ensure drug compliance, occurrence of drug-related side effects or respiratory symptoms. The final visit 4 will mark the end of study at 12 weeks from randomisation when a repeat nasopharyngeal swab for SARS-CoV-2 RT-PCR will be taken.The primary outcome measures will be prevention of SARS-CoV-2 infection as determined by a negative RT-PCR in the experimental arm at the end of 12 weeks and HCQ safety as determined by occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthcare workers all genders ≥ 18 to ≤ 60 years of age upon study consent.
* Healthcare workers (doctors and nurses) at Services hospital, Lahore considered work at high-risk of SARS-CoV-2 exposure (defined below):

  * Healthcare workers in Corona triage areas.
  * Healthcare workers in Corona Isolation Units.
  * Healthcare workers in Corona ICUs.
  * Healthcare workers in general medical wards.
  * Healthcare workers in general surgical wards.
  * Healthcare workers in other units not directly dealing with suspected Corona patients e.g. Endocrinology department
* Afebrile with no constitutional symptoms.
* No household contact with confirmed active SARS-CoV-2 infection in the last 3 weeks.
* Negative PCR at visit 0.
* Willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Willing to not take any other medicines especially fluoroquinolones and macrolides for the duration of study.
* Signed informed consent, demonstrating that the subject understands the interventions required for the study and the purpose of the study.

Exclusion Criteria:

* Participation in other investigational clinical trials for the treatment or prevention of SARS-CoV-2 infection within 30days.
* Subjects unwilling to practice at least one highly effective method of birth control for the duration of the study.
* Having a prior history of blood disorders such as aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia or prior history of glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.
* Having H/O skin disorders e.g. dermatitis, psoriasis or porphyria.
* Taking any of the following medication:

  * Anti-arrythmic agents including digoxin.
  * GI drugs including antacids, proton-pump inhibitors, cimetidine.
  * Anti-cancer treatment including methotrexate, cyclosporin.
  * Anti-diabetic agents including insulin.
  * Corticosteroids.
  * Drugs causing QT interval prolongation especially antidepressants, anti-epileptics and macrolides.
  * Drugs affecting electrolyte balance including diuretics, laxatives.
  * Drug allergies: 4-Aminoquinolines.
* Pre-existing retinopathy/maculopathy of the eye.
* Known chronic liver disease or cirrhosis, including hepatitis B and/or untreated hepatitis.
* Previous history of severe hypoglycaemia.
* Known case of renal disease.
* Untreated or uncontrolled active bacterial, fungal infection.
* Known or suspected active drug or alcohol abuse.
* Women who are pregnant or breastfeeding.
* Known hypersensitivity to any component of the study drug.
* A known history of prolonged QT syndrome or history of additional risk factors for arrythmias (e.g., heart failure, family history of Long QT Syndrome).
* Known H/O respiratory disorders e.g. asthma, chronic obstructive pulmonary disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 374 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Prevention of SARS-CoV-2 as determined by negative RT-PCR at the end of 12 week study period | From date of randomization until study completion 12 weeks after treatment initiation
  Negative RT-PCR for SARS-CoV-2 both at baseline and at end of 12 weeks in experimental arm
Safety as determined by presence or absence of any adverse event related with hydroxychloroquine treatment | From date of randomization until the appearance of symptoms or study completion 12 weeks after treatment initiation
  To assess the presence or absence of side effects from HCQ treatment.

SECONDARY OUTCOMES:
Confirmed SARS-CoV-2 infection based on symptoms and confirmed by RT-PCR | From date of randomization until the appearance of symptoms or study completion 12 weeks after treatment initiation
  Symptomatic infection by SARS-CoV-2 defined as cough, dyspnea, fever, myalgia, arthralgia or rhinorrhea.
Clinical disease severity in confirmed SARS-CoV-2 participants | From date of randomization until the appearance of symptoms or study completion 12 weeks after treatment initiation
  Disease severity including i) asymptomatic. ii) Mild symptoms but ambulatory. iii) Moderate symptoms requiring hospitalisation. iv) severe symptoms requiring ICU care and oxygen. v) Severe symptoms requiring assisted mechanical ventilation. vi) Death.
Incidence of any acute respiratory infection | From date of randomization until the appearance of symptoms or study completion 12 weeks after treatment initiation
  Symptomatic non-COVID viral infection (any other acute respiratory illness with fever but without evidence of epidemiological risk factors such as close contact with SARS-CoV-2 positive patient or travel to or residence in high-risk area).

CONTACTS AND LOCATIONS:
Overall Officials: Saira Burney, FRCP (Edin), Principal Investigator — SIMS

IPD SHARING:
Plan to Share IPD: No